CLINICAL TRIAL: NCT05421260
Title: Paediatric Spinal Cord Injury and Long-term Social Outcomes.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1 815
Record Dates: First submitted 2022-04-27; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult onset SCI: Spinal cord injury accident when the patient is over the age of 18 years old.
- Paediatric onset SCI: Spinal cord injury accident when the patient is under the age of 18 years old.

SUMMARY:
To provide the overall quality of life (QOL), activity and participation values for adults with paediatric onset spinal cord injury (SCI), stratified by injury level, neurological status and compare it with matched controls with adults with adult-onset SCI.

DETAILED DESCRIPTION:
Evidence obtained from adult studies demonstrate that SCI can be a devastating experience that may result in reduced independence and change one's ability to participate in meaningful roles and activities.

Sadly, there is a paucity of similar studies into paediatric onset SCI. The profile of paediatric patients with SCI is different from adults and their long-term wellbeing outcomes are not well researched. Maximizing activity and participation following SCI is an important aspect of rehabilitation. Community integration is a long process that might take months to years after discharge from hospital after the initial injury. After discharge from hospital the subsequent management is done by community team comprising of physio and occupational therapists who are pivotal in supporting re-engagement in social activities.

There is a need for thorough analysis regarding the social outcomes of adults living with paediatric onset SCI. Quality of life, or life satisfaction, is arguably the most important outcome for children and adolescents with SCIs. This outcome may be the key to assessing the success of our treatment pathways and will allow us to target the resources available for rehabilitation to maximize the effects of rehabilitation programs.

There are large gaps in the literature regarding paediatric SCIs. Clinicians often struggle to give informed answers to questions such as:

* Will a child with SCI experience good quality of life in adulthood?
* Is there a difference in social activity and participation between adult onset and paediatric onset injuries?
* What helps social activity and participation of SCI patients?
* Is tetraplegia worse than paraplegia for social participation?
* Does social participation affect quality of life?
* Where can we target resources in rehabilitation program?

This study aspires to address these questions by conducting this questionnaire study to understand the factors that affect social participation. This will enable to highlight areas to target future resources for rehabilitation programmes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 60 years
* SCI for over 5 years duration

Exclusion Criteria:

* Patients unable to speak and understand English
* Patients not able to speak on phone
* Patients with intellectual disability affecting their ability to speak without aids.
* Cauda equina syndrome

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult and paediatric onset SCI patients who have had their SCI for over 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
To compare long term quality of life between paediatric and adult-onset SCI patients. | This interview (a combination of these validated questionnaires) will take place within 30 days of seeking consent from the participant. Once the interview has taken place, the participant has completed the research study.
  By interviewing the participant, using a validated questionnaire from the International SCI data set, the Quality of Life basic data set, version 1.0, the long term quality of life can be assessed.
To compare long term social activity and social participation between paediatric and adult-onset SCI patients. | This interview (a combination of these validated questionnaires) will take place within 30 days of seeking consent from the participant. Once the interview has taken place, the participant has completed the research study.
  By interviewing the participant, using a validated questionnaire from the International SCI data set, Activities and participation basic data set, Version 1.0, August 2012, the social activity and social participation can be assessed.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogel LC, Betz RR, Mulcahey MJ. Spinal cord injuries in children and adolescents. Handb Clin Neurol. 2012;109:131-48. doi: 10.1016/B978-0-444-52137-8.00008-5. PMID 23098710
- [Background] Parent S, Mac-Thiong JM, Roy-Beaudry M, Sosa JF, Labelle H. Spinal cord injury in the pediatric population: a systematic review of the literature. J Neurotrauma. 2011 Aug;28(8):1515-24. doi: 10.1089/neu.2009.1153. Epub 2011 Jun 9. PMID 21501096
- [Background] Vogel L, Mulcahy MJ, Betz RR. The child with a spinal cord injury. Dev Med Child Neurol. 1997 Mar;39(3):202-7. doi: 10.1111/j.1469-8749.1997.tb07411.x. No abstract available. PMID 9112971
- [Background] Vogel LC, Klaas SJ, Lubicky JP, Anderson CJ. Long-term outcomes and life satisfaction of adults who had pediatric spinal cord injuries. Arch Phys Med Rehabil. 1998 Dec;79(12):1496-503. doi: 10.1016/s0003-9993(98)90409-9. PMID 9862289
- [Background] Kulshrestha R, Kumar N, Chowdhury JR, Osman A, El Masri W. Long-term outcome of paediatric spinal cord injury. Trauma, 2017, 19,1_suppl: 75-82.
- [Background] Post MW, van Leeuwen CM. Psychosocial issues in spinal cord injury: a review. Spinal Cord. 2012 May;50(5):382-9. doi: 10.1038/sc.2011.182. Epub 2012 Jan 24. PMID 22270190
- [Background] Barclay L, Lentin P, Bourke-Taylor H, McDonald R. The experiences of social and community participation of people with non-traumatic spinal cord injury. Aust Occup Ther J. 2019 Feb;66(1):61-67. doi: 10.1111/1440-1630.12522. Epub 2018 Aug 29. PMID 30156293
- [Background] Barclay L, Callaway L, McDonald R, Farnworth L, Brown T, Broom L. Time Use following Spinal Cord Injury: An Examination of the Literature. British Journal of Occupational Therapy. 2011; 74 (12): 573-580
- [Background] Biering-Sorensen F, Charlifue S, DeVivo M, Noonan V, Post M, Stripling T, Wing P. International Spinal Cord Injury Data Sets. Spinal Cord. 2006 Sep;44(9):530-4. doi: 10.1038/sj.sc.3101930. PMID 16955072